CLINICAL TRIAL: NCT01939067
Title: Pulmonary Mechanics in Preterm Infants Treated With Heated Humidified High Flow Nasal Cannula as Compared to Nasal Continuous Positive Airway Pressure.
Brief Title: Infant Pulmonary Mechanics: High Flow Nasal Cannula Versus Nasal CPAP
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Application for regulatory approval withdrawn
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-009882
Record Dates: First submitted 2013-08-30; First posted 2013-09-11 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Respiratory Distress; Lung Injury
Keywords: respiratory distress; Heated Humidified High Flow Nasal Cannula (HHHFNC); HHHFNC; noninvasive nasal continuous positive airway pressure (NCPAP); NCPAP
MeSH Terms: conditions — Dyspnea; Lung Injury | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HHHFNC (Other): Treatment of respiratory distress by Heated Humidified High Flow Nasal Cannula (HHHFNC).
  Escalation of the ventilatory support per protocol and the attending physician.
  Interventions: Device: Heated Humidified High Flow Nasal Cannula
- NCPAP (Other): Treatment of respiratory distress by nasal continuous positive airway pressure (NCPAP).
  Escalation of the ventilatory support per protocol and the attending physician.
  Interventions: Device: Nasal Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Heated Humidified High Flow Nasal Cannula — Biweekly measurement of lung mechanics (dynamic compliance, airway resistance, work of breathing) and chest wall asynchrony measures while on HHHFNC and weekly when weaned off until 40 weeks post conceptional age or discharge. Recording of the level and the type of respiratory support and all cross over respiratory support devices. Recording of all growth parameters, neonatal morbidities and therapies.
  Arms: HHHFNC
Device: Nasal Continuous Positive Airway Pressure — Biweekly measurement of lung mechanics (dynamic compliance, airway resistance, work of breathing) and chest wall asynchrony measures while on NCPAP and weekly when weaned off until 40 weeks post conceptional age or discharge. Recording of the level and the type of respiratory support and all cross over respiratory support devices. Recording of all growth parameters, neonatal morbidities and therapies.
  Arms: NCPAP

SUMMARY:
This study is designed to evaluate the effect of heated humidified high flow nasal cannula (HHHFNC) as compared to noninvasive nasal continuous positive airway pressure (NCPAP) on lung function as a measure of lung injury in preterm infants born at 28 to 37 weeks gestation requiring continuing respiratory support.

DETAILED DESCRIPTION:
Respiratory distress and the need for respiratory support continues to be a common problem for preterm infants. Presence of the breathing tube and duration of respirator provided breaths have been shown to be associated with increased risk for secondary lung injury and subsequent development of chronic lung disease of prematurity. Early application of noninvasive nasal continuous positive airway pressure (NCPAP) has been shown to be an effective, non-invasive, mode of respiratory support in preterm infants and to be associated with a lower incidence of chronic lung disease. A recently published large randomized multicenter study concluded that, among infants born at 28 weeks and longer gestation, heated humidified high flow nasal cannula (HHHFNC) had similar clinical efficacy and safety as compared to NCPAP. Both NCPAP and HHHFNC are currently used to assist infants with breathing problems.

This study is designed to evaluate the effect of HHHFNC as compared to NCPAP on lung function as a measure of lung injury in preterm infants born at 28 to 37 weeks gestation requiring continuing respiratory support. In this study, infants will remain on the assigned treatment of either NCPAP or HHHFNC until they require more support as provided by a respirator or until a treatment cross-over from NCPAP to HHHFNC, or the reverse, as decided by their attending physician. The infant's respiratory support will be managed according to his/her attending doctor as per accepted standards of care. A pulmonary function test will be performed twice weekly on each enrolled infant while receiving either NCPAP or HHHFNC support, followed-up by once weekly lung function measurements post respiratory support while infants are breathing only room air until discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight greater than or equal to 1000 grams.
2. Gestational age at birth between 28 weeks and 37 weeks (28 0/7 to 37 6/7 weeks inclusive).
3. Candidate for non-invasive respiratory support as a result of:

   1. An intention to manage the infant with non-invasive (no endotracheal tube) respiratory support.
   2. An intention to extubate an infant being managed with intubated respiratory support to non-invasive respiratory support.
4. Subjects must have a guardian or acceptable surrogate capable of giving consent on his/her behalf.

Exclusion Criteria:

1. Birth weight less than 1000 grams.
2. Estimated gestation at birth less than 28 weeks or greater than 37 6/7 weeks.
3. Active air leak syndrome.
4. Subjects will not be eligible if they are not considered viable.
5. Infants with abnormalities of the upper and lower airways
6. Infants with significant abdominal or respiratory malformations .

Ages: 2 Hours to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary mechanics and chest wall asynchrony measures. | 2 years
  Pulmonary mechanics measures consisting of dynamic lung compliance, airway resistance, and work of breathing and chest wall asynchrony measures consisting of thoracoabdominal asynchrony, labored breathing index and rib cage to abdominal phase relation during the total breath are measured in preterm infants treated with HHHFNC and compared to the same measurements in preterm infants treated with NCPAP.

SECONDARY OUTCOMES:
Duration of respiratory support or oxygen use up to the time of discharge from the NICU. | 2 years
  The total number of days while infants are on any type of respiratory support or oxygen use prior to discharge in preterm infants treated with HHHFNC compared to NCPAP during their hospital stay.
The incidence of potential adverse outcomes associated with HHHFNC or NCPAP. | 2 years
  The number and percentage of infants in each group with adverse effects such as facial and upper airways injury associated with the use of HHHFNC or NCPAP.
Time needed to establish full enteral feeds | 2 years
  The total number of days needed to establish full enteral feeds in preterm infants treated with HHHFNC as compared to preterm infants treated with NCPAP.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Abbasi, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States